CLINICAL TRIAL: NCT07361484
Title: A Global, Multicenter, Randomized, Double-blinded, Phase 3 Study of Docetaxel + Plinabulin Compared to Docetaxel + Placebo in Patients With Advanced or Metastatic Non-squamous Non-Small Cell Lung Cancer With EGFR, ALK, ROS, and RET Wild Type After Progressing on Prior Immunotherapy (Anti-PD-1/L1 Antibody) and Platinum-based Chemotherapy (DUBLIN-4)
Brief Title: Docetaxel Plus Plinabulin vs Docetaxel Plus Placebo in Advanced/Metastatic Non-Squamous NSCLC After PD-1/PD-L1 Therapy and Platinum Chemotherapy (DUBLIN-4)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeyondSpring Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPI 2358 112
Record Dates: First submitted 2026-01-19; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer; Non-squamous Non-Small Cell Lung Cance
Keywords: Advanced NSCLC; Metastatic NSCLC; Non-squamous NSCLC; EGFR wild type; ALK wild type; ROS1 wild type; RET wild type; Docetaxel; Plinabulin; BPI-2358; DUBLIN-4
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — NPI 2358; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Docetaxel + Plinabulin (Experimental): Participants will receive docetaxel IV infusion on Day 1 of each 21-day cycle plus plinabulin IV infusion on Days 1 and 8. Treatment continues until disease progression, unacceptable toxicity, death, withdrawal, or sponsor/investigator decision.
  Interventions: Drug: Plinabulin; Drug: Docetaxel
- Docetaxel + Placebo (Placebo Comparator): Participants will receive docetaxel IV infusion on Day 1 of each 21-day cycle plus matching placebo IV infusion on Days 1 and 8. Treatment continues until disease progression, unacceptable toxicity, death, withdrawal, or sponsor/investigator decision.
  Interventions: Drug: Docetaxel; Drug: Placebo (matching plinabulin placebo)

INTERVENTIONS:
Drug: Plinabulin — Plinabulin will be administered by IV infusion at 30 mg/m² over approximately 1 hour on Days 1 and 8 of each 21-day treatment cycle. On Day 1, plinabulin will be administered approximately 1 hour after completion of the docetaxel infusion.
  Arms: Docetaxel + Plinabulin
Drug: Docetaxel — Docetaxel will be administered by intravenous (IV) infusion at 75 mg/m² over approximately 1 hour on Day 1 of each 21-day treatment cycle.
Drug: Placebo (matching plinabulin placebo) — Matching placebo will be administered by IV infusion over approximately 1 hour on Days 1 and 8 of each 21-day treatment cycle. On Day 1, placebo will be administered approximately 1 hour after completion of the docetaxel infusion.
  Arms: Docetaxel + Placebo

SUMMARY:
This is a global, multicenter, randomized, double-blind, placebo-controlled Phase 3 study evaluating docetaxel plus plinabulin versus docetaxel plus placebo in participants with advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) without EGFR, ALK, ROS1, or RET alterations who have experienced disease progression after prior anti-PD-1/PD-L1 immunotherapy and platinum-based chemotherapy. Approximately 442 participants will be randomized 1:1 to receive docetaxel (75 mg/m² IV on Day 1 of each 21-day cycle) in combination with plinabulin (30 mg/m² IV on Days 1 and 8) or matching placebo. Treatment will continue until disease progression, unacceptable toxicity, death, withdrawal of consent, or sponsor/investigator decision. Tumor assessments will be performed regularly per RECIST v1.1, and participants will be followed for survival after treatment discontinuation. The primary objective is to compare overall survival between treatment arms; secondary objectives include evaluation of progression-free survival, objective response rate, duration of response, disease control, incidence of Grade 4 neutropenia, quality of life, and safety/tolerability.

DETAILED DESCRIPTION:
Participants with advanced or metastatic non-squamous non-small cell lung cancer (NSCLC) who have progressed following prior anti-PD-1/PD-L1 immunotherapy and platinum-based chemotherapy have limited treatment options and docetaxel remains a commonly used standard therapy in this setting. Plinabulin is a first-in-class small molecule with a distinct mechanism that may enhance anti-tumor activity and may mitigate chemotherapy-associated neutropenia. This study (DUBLIN-4) is designed to evaluate whether the addition of plinabulin to docetaxel improves clinical outcomes compared with docetaxel alone in this post-immunotherapy and post-platinum population without EGFR, ALK, ROS1, or RET alterations.

This is a global, multicenter, randomized, double-blind, placebo-controlled Phase 3 study. Participants will be randomized in a 1:1 ratio to receive docetaxel in combination with plinabulin or matching placebo. Randomization will be stratified by geographic region (Asian countries vs Western countries), current line of therapy (2nd vs 3rd line), and prior progression-free survival duration on PD-1/PD-L1 inhibitor therapy (≥6 months vs <6 months).

Efficacy will be evaluated using standard radiographic tumor assessments and response criteria, with additional evaluation of clinically relevant outcomes in this treatment setting, including overall survival, progression-free survival, and objective response. Safety will be assessed throughout the study by monitoring adverse events, laboratory parameters, and other routine clinical assessments. The study also includes evaluation of patient-reported quality of life and the incidence of severe neutropenia as an important tolerability endpoint for docetaxel-based treatment.

Participants who discontinue study treatment will enter follow-up, including a safety follow-up after treatment discontinuation and ongoing survival follow-up. Sparse pharmacokinetic samples will be collected to support population pharmacokinetic analyses of plinabulin.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 18 years of age or older at the time of signing the ICF
2. Willing and able to sign an ICF;
3. Non-squamous NSCLC with EGFR, ALK, ROS and RET wild type who have been diagnosed by histopathological and/or cytological examination as being ineligible for surgical treatment and have locally advanced (stage IIIb) or metastatic (stage IV) diseases, or have recurrent and progressive disease after local treatment (if there are multiple tumor components, classify the main cell type):

   * Developed disease progression after treatment with PD-1/L1 inhibitors and platinum-based chemotherapy in advanced non-squamous NSCLC with EGFR, ALK, ROS and RET wild type
   * Treatment progression with anti-PD-1/L1 inhibitors and platinum-based chemotherapy administered either concurrently or sequentially as part of the same first-line treatment plan, or as two separate prior lines of systemic therapy, (does not count preoperative and adjuvant therapy) is defined to meet all of the following criteria:

     1. Demonstrated disease progression after anti-PD-1/L1 and platinum-based chemotherapy concurrently or sequentially as defined by RECIST v1.1
     2. Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression. The disease progression to the first administration of the IMP should not exceed 60 days
     3. Achieved PFS of anti- PD-1/L1 treatment for at least 3 months
4. ECOG performance status of 0 to 1
5. All AEs from any previous systemic therapy, surgery or radiotherapy must have been resolved to CTCAE v5.0 Grade ≤1 or baseline
6. Adequate organ function, within 7 days prior to administration of the IMP by the local laboratory:

   * Hemoglobin ≥9 g/dL independent of transfusions or growth factor support
   * ANC ≥1.5×109/L independent of growth factor support
   * Platelet count ≥100×109/L independent of blood transfusion
   * Serum total bilirubin ≤ the ULN, unless the participant has a diagnosis of Gilbert's disease in which case serum total bilirubin ≤3.0×ULN
   * AST and ALT ≤2.5×ULN (≤1.5×ULN if alkaline phosphatase is >2.5× ULN, ≤5xULN with liver metastasis)
   * CrCl ≥50 mL/min (as calculated by the Cockcroft-Gault formula)
7. Life expectancy of at least 3 months
8. Female participants of childbearing potential have a negative pregnancy test at baseline. Females of childbearing potential are defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti estrogens, or ovarian suppression
9. Female participants must be in a non-pregnant and non-lactating state, and females of childbearing potential (including their partners) are willing to voluntarily adopt effective contraceptive measures from the screening period until 3 months after the last administration of the IMP. Females of childbearing potential (ie, menstruating women) must have a negative urine pregnancy test (positive urine tests are to be confirmed by serum test) documented within the 24-hour period prior to the first dose of IMP

   * Sexually active females of childbearing potential enrolled in the study must agree to use 2 forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of IMP. Effective birth control includes: (a) intrauterine device plus 1 barrier method; (b) on stable doses of hormonal contraception for at least 3 months (eg, oral, injectable, implant, transdermal) plus 1 barrier method; (c) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm); or (d) a vasectomized partner
   * Male participants who are sexually active and who are partners of pre menopausal women must agree to use 2 forms of accepted contraception during the treatment period and for at least 3 months after the last dose of IMP

Exclusion Criteria:

1. Administration of chemotherapy, immunotherapy, biotherapy, targeted, or radiation therapy or investigational agent (therapeutic or diagnostic) within 3 weeks prior to the first dose of IMP. Major surgery, other than diagnostic surgery, within 4 weeks before first IMP administration is exclusionary
2. Receipt of more than two prior lines of systemic anticancer therapy for locally advanced or metastatic non-small cell lung cancer. Neoadjuvant and adjuvant systemic therapies are not counted as prior lines of therapy
3. Any of the following cardiac criteria experienced currently or within the last 6 months:

   * Congestive heart failure (New York Heart Association ≥Class 2)
   * Any clinically significant abnormalities (as assessed by the investigator) in rhythm, conduction, or morphology of resting ECGs, eg, complete left bundle branch block or third-degree heart block
   * Acute coronary syndrome
   * Clinically significant uncontrolled cardiac arrhythmia
4. Any of the following cardiac criteria experienced currently:

   * Mean QTC interval corrected (Friderica) >470 ms
   * Left ventricular ejection fraction <50% or the lower limit of normal (per institutional standard)
5. Evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension (>160 mmHg systolic and 100 mmHg diastolic in spite of anti hypertension medication), uncontrolled diabetes mellitus, active bleeding diatheses, as determined by the investigator
6. Participants who have received prior treatment with docetaxel
7. Prior transient ischemic attack or cerebrovascular accident within the past year
8. History of hemorrhagic diarrhea, inflammatory bowel disease or active uncontrolled peptic ulcer disease (concomitant therapy with ranitidine or its equivalent and/or omeprazole or its equivalent is acceptable). History of ileus or other significant gastrointestinal disorder known to predispose to ileus or chronic bowel hypomotility
9. Active bacterial, viral, or fungal infection requiring systemic therapy
10. A current or a known history of acquired immunodeficiency syndrome-defining illness, or HIV infection with a CD4+ T-cell count <350 cells/µL and an HIV viral load more than 400 copies/µL
11. Participants with active viral (any etiology) hepatitis are excluded. However, participants with serologic evidence of chronic HBV infection (defined by a positive hepatitis B surface antigen test and a positive anti-hepatitis core antigen antibody test) who have a viral load below the limit quantification (HBV DNA titer <1000 cps/mL or 200 IU/mL), and are not currently on viral suppressive therapy may be eligible and should be discussed with the medical monitor. Participants with a history of hepatitis C virus infection who have completed curative antiviral treatment and have a viral load below the limit of quantitation may be eligible and should be discussed with the medical monitor
12. Known prior hypersensitivity reaction to any product containing polysorbate 80, polyoxyethylene 15-hydroxystearate/macrogol 15-hydroxystearate (Solutol HS 15/Kolliphor HS 15), and docetaxel
13. Other malignancies, unless in remission for >3 years (non-melanoma skin cancer or carcinoma in situ of the cervix treated with curative intent is not exclusionary)
14. Participants with central nervous system metastasis with hemorrhagic features and symptomatic brain metastases uncontrolled by a stable dose of steroids (≤4 mg dexamethasone or equivalent)
15. Participants with brain radiation within 7 days before screening
16. Participants with leptomeningeal diseases
17. History or evidence of any other clinically significant condition or disease (with the exception of those outlined above) that, in the opinion of the investigator, would be a risk to participant safety or interfere with the study evaluation, procedures or completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Approximately 2 years after study initiation.
  OS is defined as the time from randomization to death from any cause

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Approximately 2 years after study initiation.
  Time from randomization to the first documentation of disease progression per RECIST v1.1 or death from any cause, whichever occurs first.
Objective Response Rate (ORR) | Approximately 2 years after study initiation.
  Proportion of participants with best overall response of complete response (CR) or partial response (PR) per RECIST v1.1.
Incidence of Grade 4 Neutropenia (Cycle 1 Day 8 ANC) | At Day 8 of Cycle 1 (approximately 1 week after the first dose; each treatment cycle is 21 days).
  Proportion of participants with Grade 4 neutropenia, defined as absolute neutrophil count (ANC) <0.5 × 10^9/L, based on ANC on Day 8 of Cycle 1.
Overall Survival (OS) Rate at Month 24 | 24 months after randomization.
  Proportion of participants alive at 24 months after randomization.
Overall Survival (OS) Rate at Month 36 | 36 months after randomization.
  Proportion of participants alive at 36 months after randomization.
Duration of Response (DoR) | Approximately 2 years after study initiation.
  Time from first documented CR or PR (whichever occurs first) until disease progression per RECIST v1.1 or death from any cause.
Disease Control Rate (DCR) | Approximately 2 years after study initiation.
  Proportion of participants with CR, PR, or stable disease (SD) lasting ≥6 months per RECIST v1.1.
Incidence of New Brain Metastases | Approximately 2 years after study initiation.
  Incidence of new brain metastases based on brain imaging (MRI or head CT).
Quality of Life (QoL) - EORTC QLQ-LC13 | Approximately 2 years after study initiation.
  Change from baseline in EORTC QLQ-LC13 scores. Quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Lung Cancer 13 (EORTC QLQ-LC13). Scores are transformed to a 0 to 100 scale. Higher scores indicate worse symptoms / greater symptom burden (worse outcome).
Incidence and Severity of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Approximately 2 years after study initiation.
  TEAEs and SAEs will be assessed throughout the study and summarized by frequency, severity (per CTCAE), and relationship to study treatment.

OTHER OUTCOMES:
Metastasis-Free Survival (MFS) | Approximately 2 years after study initiation.
  MFS is defined as the time from randomization to the first occurrence of new distant metastasis or death from any cause, whichever occurs first.

REFERENCES:
- See also: BEYONDSPRING PHARMACEUTICALS, INC. WEBSITE — https://beyondspringpharma.com/